CLINICAL TRIAL: NCT04414553
Title: Community Active and Healthy Families: Family-Centered Obesity Treatment for Latino Children
Brief Title: Community Active and Healthy Families
Acronym: CommunityAHF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-1337
Record Dates: First submitted 2020-05-20; First posted 2020-06-04 (Actual); Results first posted 2025-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Obesity, Childhood
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Intervention Model Description: Pre/Post
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Community-AHF (Experimental): Participants in this arm will receive the Community Active and Healthy Families Intervention
  Interventions: Behavioral: Community Active and Healthy Families

INTERVENTIONS:
Behavioral: Community Active and Healthy Families — Community-AHF will consist of eight, semimonthly 2-hour group appointments. Community-AHF sessions will target two areas: 1) Practical information regarding importance of healthy behaviors, and 2) Problem-solving skills to overcome barriers to improving diet and increasing physical activity and other related healthy behaviors. Each session covers specific objectives, includes a number of complementary activities and provides participants with take-home materials to facilitate behavior change.
  Community-AHF will be delivered by a nurse and a Community Health Worker (CHW) trained by a consultant nutritionist and study investigators. The CHW will contact families between group sessions to discuss challenges and successes regarding lifestyle changes.

SUMMARY:
To address childhood overweight disparities among Latino children in immigrant families a pilot trial of a community-based obesity treatment program, Community Active and Healthy Families (AHF), among 5-12 year old overweight and obese Latino children in immigrant families using pre/post design will be conducted.

The hypothesis is that children participating in Community-AHF will demonstrate a reduction in child body mass index as measured by %BMIp95 (primary outcome) and improved diet physical activity behaviors (secondary outcomes) at intervention completion compared with pre-intervention

DETAILED DESCRIPTION:
To address childhood overweight disparities among Latino children in immigrant families a pilot trial of a community-based obesity treatment program, Community Active and Healthy Families (AHF), among 5-12 year old overweight and obese Latino children in immigrant families using a pre/post design will be conducted.

As this is a pilot study, the study will not be powered to detect statistically significant differences pre- and post- intervention. The investigators will measure the average change in %BMIp95 between baseline and completion of the Community-AHF active phase. Without a counterfactual (control group) the investigators will not be able assign responsibility to Community-AHF for any observed improvements. Change in %BMIp95 across the study period will provide data to test our hypotheses and will inform statistical power analyses for a subsequent trial. This pre- and post-intervention data is ideal for generating sample size estimates for a larger randomized control trial in the same population.

The investigators will conduct within-individual analyses for each outcome of interest. The investigators will only analyze participants who contribute pre and post measures in order to avoid biases that can occur when analyses are conducted with all available data. For each outcome for which a participant contributes pre and post measurements, the investigators will calculate pre and post means, standard deviations, differences in means and the p-value of the difference. The investigators will conduct preliminary analyses of outcomes according to subgroups defined by rate of attendance at intervention sessions. If adequate data are available, the investigators will explore the possibility of a nonresponse analysis.

ELIGIBILITY:
Inclusion Criteria:

* Child age 5-12 years with Parent/Caregiver age of 18 or more years
* Child BMI >/= 85th percentile for age
* Parent is foreign-born, self identifies as Latino/Hispanic and speaks Spanish
* Parental commitment to participate in a 4-month intervention

Exclusion Criteria:

* Child health condition that prevents diet modification or engaging in physical activity
* Child BMI >40kg/m2

Ages: 5 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2023-03-13 (Actual); Primary Completion 2023-09-23 (Actual); Study Completion 2023-11-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa R DeCamp, MD, MSPH, Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - University of Colorado, Aurora, Colorado
  - Johns Hopkins University, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No
Pending further study planning we will make this decision.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participating families were recruited via referral from their primary care provider at academic-based general pediatrics clinics (both sites) or community-based recruitment from among participants in programming at a Latino immigrant-serving family resource center and at nearby elementary schools. (Colorado only). Recruitment occurred between Jan-March 2023.
Pre-assignment Details: This was a single arm study where all participants who enrolled were assigned to complete the study intervention.
Groups:
- Community-AHF: Participants in this arm will receive the Community Active and Healthy Families Intervention
  Community Active and Healthy Families: Community-AHF will consist of eight, semimonthly 2-hour group appointments. Community-AHF sessions will target two areas: 1) Practical information regarding importance of healthy behaviors, and 2) Problem-solving skills to overcome barriers to improving diet and increasing physical activity and other related healthy behaviors. Each session covers specific objectives, includes a number of complementary activities and provides participants with take-home materials to facilitate behavior change.
  Community-AHF will be delivered by a nurse and a Community Health Worker (CHW) trained by a consultant nutritionist and study investigators. The CHW will contact families between group sessions to discuss challenges and successes regarding lifestyle changes.
Period: Overall Study
Arm/Group | Community-AHF
Started | 78
# of Parents | 39
# of Children | 39
Completed (these 58 participants include 29 parents and 29 children) | 58
Not Completed | 20
Not completed — Lost to Follow-up | 20

BASELINE CHARACTERISTICS:
Population: The baseline analyses describe the 39 dyads that participate in the Community AHF Pilot.
Arm/Group | Community-AHF
Number analyzed (Participants) | 78
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 39
  Between 18 and 65 years | 39
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Mean Child and Parent Age as separate categories Population: The # analyzed per row differs as we are looking at parent and child mean age separately
  years
    Child Age: number analyzed (Participants) | 39
    Child Age | 10.1 (2.2)
    Parent Age: number analyzed (Participants) | 39
    Parent Age | 39.6 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54
  Male | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Latino Ethnicity of any race | 78
Region of Enrollment [Number; unit: participants]
  United States | 78
Pre-program %BMIp95, mean (SD) [Mean (Standard Deviation); unit: percent] — Our primary outcome age- and sex-specific BMI expressed as percent of the 95th percentile (%BMIp95) based on Centers for Disease Control's 2000 growth charts. %BMIp95 is recommended in longitudinal studies due to constraints of BMI z-scores among children with severe obesity. Population: This outcome only applies to the child participant
  percent
    number analyzed (Participants) | 39
    (all) | 125.35 (23.11)
BMI Category [Count of Participants; unit: Participants] — Ths describes the category of overweight/obesity where the child measured at baseline Population: Only children had BMI outcomes measured
  Participants
    number analyzed (Participants) | 39
    Overweight (BMI 85-94%tile) | 1
    Obese (BMI 95-99%tile) | 2
    Severe obesity (BMI >99%tile) | 36
Child Physical Activity [Number; unit: participants] — # of days per week the child is physically active Population: This measure of physical activity in the last week applies to the child only
  participants
    Low Health Risk (6-7 days/week): number analyzed (Participants) | 39
    Low Health Risk (6-7 days/week) | 5
    Medium Health Risk (3-5 days/week) | 11
    High Health Risk (0-1 times/week) | 23
    Medical Contraindication | 0
Parent Self Efficacy [Mean (Standard Deviation); unit: units on a scale] — Parent Self-Efficacy for Healthy Weight Promotion Population: This measure is only for the parents
  units on a scale
    number analyzed (Participants) | 39
    (all) | 21.00 (1.87)
Parent Perceived Stress [Mean (Standard Deviation); unit: units on a scale] — The measure is a parent self report of stress using the validated Perceived Stress Scale-10 Population: This is a parent only measure
  units on a scale
    number analyzed (Participants) | 39
    (all) | 18.10 (20.52)

OUTCOME MEASURES:

1. Primary Outcome: %BMIp95
Description: Age- and sex-specific BMI expressed as percent of the 95th percentile. Child Body Mass Index is calculated from child height and weight measurement.
Time Frame: 4 months
Population: Children who had both pre/post program data
Measure: Mean (Standard Deviation); unit: percent of the 95th percentile of BMI
Arm/Group | Community-AHF
Number analyzed (Participants) | 29
percent of the 95th percentile of BMI | 122.35 (15.95)
Statistical Analysis 1: Comparison: Community-AHF; This compares pre/post data; Test type: Superiority; p = 0.29, t-test, 2 sided — Threshold for statistical significance was <0.05

2. Primary Outcome: BMI Category
Description: This measure examines BMI category of overweight, obesity, severe obesity pre/post program
Time Frame: 4 months
Population: Children with complete pre/post data
Measure: Count of Participants; unit: Participants
Arm/Group | Community-AHF
Number analyzed (Participants) | 29
Participants
  Overweight (BMI 85-94%tile) | 0
  Obese (BMI 95-99%tile) | 3
  Severe obesity (BMI >99%tile) | 26
Statistical Analysis 1: Comparison: Community-AHF; Test type: Superiority; p = 0.35, Chi-squared

3. Secondary Outcome: Child Physical Activity
Description: parent-report of the number of days the child is physically active for 60 minutes during a typical week Range 0-7, Higher scores indicate a better outcome (more physical activity)
Time Frame: 4months
Population: Participants with complete pre/post data
Measure: Count of Participants; unit: Participants
Arm/Group | Community-AHF
Number analyzed (Participants) | 29
Participants
  Low Health Risk (6-7 days/week) | 13
  Medium Health Risk (3-5 days/week) | 5
  Low Health Risk (0-1 days/week) | 10
  Medical Contraindication | 1
Statistical Analysis 1: Comparison: Community-AHF; Test type: Superiority; p = 0.21, Chi-squared

4. Secondary Outcome: Parenting Self-Efficacy
Description: 4 questions related to self efficacy Range 5-25, Higher scores indicate a better outcome (more parenting self efficacy)
Time Frame: 4 months
Population: Participants with complete pre/post data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Community-AHF
Number analyzed (Participants) | 29
units on a scale | 20.14 (1.27)
Statistical Analysis 1: Comparison: Community-AHF; Test type: Superiority; p = 0.018, t-test, 2 sided

5. Secondary Outcome: Parent Perceived Stress
Description: The 10-item Perceived Stress Score measures global perceived stress experienced across the past 30 days.
  Range: 0-40, lower scores indicate a better outcome (less stress)
Time Frame: 4 months
Population: Participants with complete pre/post data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Community-AHF
Number analyzed (Participants) | 29
units on a scale | 20.52 (6.29)
Statistical Analysis 1: Comparison: Community-AHF; Test type: Superiority; p = 0.062, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Community-AHF
All-Cause Mortality (participants affected / at risk) | 0/78
Serious Adverse Events (participants affected / at risk) | 0/78
Other Adverse Events (participants affected / at risk) | 0/78

LIMITATIONS AND CAVEATS:
This is a pilot study which is not intended to evaluate effectiveness. In addition the study had a 74% completion rate. Missing follow up data may bias the results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-13): https://cdn.clinicaltrials.gov/large-docs/53/NCT04414553/Prot_SAP_000.pdf